CLINICAL TRIAL: NCT02031458
Title: A Phase II, Multicenter, Single-Arm Study OF Atezolizumab In Patients With PD-L1-Positive Locally Advanced Or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab in Participants With Programmed Death - Ligand 1 (PD-L1) Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: BIRCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO28754; 2013-003330-32 (EudraCT Number)
Record Dates: First submitted 2013-12-16; First posted 2014-01-09 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

ARMS (1):
- Atezolizumab (Experimental)
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg IV every 3 weeks

SUMMARY:
This multicenter, single-arm study will evaluate the efficacy and safety of Atezolizumab in participants with PD-L1-positive locally advanced or metastatic non-small cell lung cancer (NSCLC). Participants will receive Atezolizumab 1200 milligrams (mg) intravenously every 3 weeks as long as participants are experiencing clinical benefit as assessed by the investigator, that is , in the absence of unacceptable toxicity or symptomatic deterioration attributed to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants greater than or equal to 18 years of age
* Locally advanced or metastatic (Stage IIIB, Stage IV, or recurrent) NSCLC
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens
* PD-L1-positive tumor status as determined by an immunohistochemistry (IHC) assay based on PD-L1 expression on tumor infiltrating immune cells and/or tumor cells performed by a central laboratory
* Measurable disease, as defined by RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Any approved anti-cancer therapy, including chemotherapy, or hormonal therapy within 3 weeks prior to initiation of study treatment; the following exception are allowed:

Hormone-replacement therapy or oral contraceptives tyrosine-kinase inhibitors (TKIs) approved for treatment of NSCLC discontinued >7 days prior to Cycle 1, Day 1

* Central nervous system (CNS) disease, including treated brain metastases
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with negligible risk of metastases or death and treated with expected curative outcome
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis (including pneumonia), drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening CT scan. History of radiation pneumonitis in the radiation field (fibrosis) id permitted
* Active hepatitis B or hepatitis C
* Human Immunodeficiency virus (HIV) positive
* Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2014-01-22 (Actual); Primary Completion 2015-05-28 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (110):
- United States (37):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - HonorHealth Research Institute - Bisgrove, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Angeles Clinic & Rsch Inst, Los Angeles, California
  - City of Hope National Medical Group, South Pasadena, California
  - Stanford Cancer Center, Stanford, California
  - University of Colorado Health Science Center; Biomedical Research Bldg. Room 511, Aurora, Colorado
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists; SCRI, Fort Myers, Florida
  - Florida Hospital Cancer Inst, Orlando, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists., St. Petersburg, Florida
  - Emory Uni - Winship Cancer Center; Hematology/Oncology, Atlanta, Georgia
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Northwestern University; Robert H. Lurie Comp Can Ctr, Chicago, Illinois
  - University Of Chicago Medical Center; Section Of Hematology/Oncology, Chicago, Illinois
  - Uni of Maryland; Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr; Hem/Onc, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Monter Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolina BioOncology Institute, PLCC, Huntersville, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University; B406 Starling-Loving Hall, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center; Hematology/Oncology, Philadelphia, Pennsylvania
  - Tennessee Oncology PLLC - Nashville (20th Ave), Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute; University of Utah, Salt Lake City, Utah
  - University of Virginia; Office of Sponsored Programs, Charlottesville, Virginia
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (5):
  - Royal North Shore Hospital; Oncology, St Leonards, New South Wales
  - Princess AleXandra Hospital; Department of Medical Oncology, Woolloongabba, Queensland
  - Austin Health, Heidelberg, Victoria
  - Peter Maccallum Cancer Institute; Medical Oncology, Melbourne, Victoria
  - Sir Charles Gairdner Hospital; Medical Oncology, Nedlands, Western Australia
- Belgium (4):
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Saint-Joseph, Charleroi
  - UZ Leuven Gasthuisberg, Leuven
  - Sint Augustinus Wilrijk, Wilrijk
- Bosnia and Herzegovina (3):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - University Clinical Center Sarajevo;Clinic for Pulmonary disease, Sarajevo
  - University Clinical Center Sarajevo;Institute of oncology, Sarajevo
- Bulgaria (2):
  - Complex Oncology Center (COC)-Plovidiv, Plovdiv
  - Specialized Hospital for Active Treatment of Oncology, Sofia
- Canada (5):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
- France (8):
  - Hopital Augustin Morvan; Oncologie Thoracique, Brest
  - Hopital Cote De Nacre; Pneumologie, Caen
  - CHU Limoges - Dupuytren; Oncologie Thoracique Cutanee, Limoges
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Hopital Arnaud De Villeneuve; Maladies Respiratoires, Montpellier
  - Centre René Gauducheau - cancer Nantes - Atlantique; Service Oncologie Médicale, Nantes
  - Nouvel Hopital Civil; Pneumologie, Strasbourg
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Georgia (4):
  - Research institute for Clinical Medicine, Tbilisi
  - Cancer Research Centre, Tbilisi
  - MediClab Georgia, Tbilisi
  - Chemotherapy and Immunotherapy Clinic Medulla, Tbilisi
- Germany (5):
  - Universitätsklinikum Essen; Innere Klinik und Poliklinik für Tumorforschung, Essen
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Klinikum Nuernberg Nord; Medizinische Klinik 3, Schwerpunkt Pneumologie, Allergologie, Schlafmedizin, Nuremberg
  - Pius-Hospital; Klinik fuer Haematologie und Onkologie, Oldenburg
  - Schwarzwald-Baar Klinikum/VS GmbH; Onkologie/Hämatologie/Infektologie, Villingen-Schwenningen
- Hong Kong (3):
  - Queen Elizabeth Hospital; Clinical Oncology, Hong Kong
  - Queen Mary Hospital; Dept. of Clinical Oncology, Hong Kong
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- Italy (3):
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 1, Milan, Lombardy
  - Az. Osp. S. Luigi Gonzaga; Malattie Apparato Respiratorio 5 Ad Indirizzo Oncologico, Orbassano, Piedmont
- Japan (11):
  - National Hospital Organization Kyushu Medical Center; Respiratory Internal Medicine, Fukuoka
  - Kanagawa Cardiovascular and Respiratory Center; Respiratory Medicine, Kanagawa
  - Yokohama Municipal Citizen'S Hospital; Respiratory Medicine, Kanagawa
  - Kitasato University Hospital; Respiratory Medicine, Kanagawa
  - Kyoto University Hospital, Respiratory Medicine, Kyoto
  - Sendai Kousei Hospital; Pulmonary Medicine, Miyagi
  - Osaka International Cancer Institute; Thoracic Oncology, Osaka
  - Kansai Medical university Hospital; Thoracic Oncology, Osaka
  - Osaka Habikino Medical Center, Osaka
  - National Cancer Center Hospital; Thoracic Medical Oncology, Tokyo
  - Toranomon Hospital; Respiratory Medicine, Tokyo
- Netherlands (3):
  - Antoni Van Leeuwenhoek Ziekenhuis; Thoracic Oncology, Amsterdam
  - Amphia Ziekenhuis; Afdeling Longziekten, Breda
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
- Singapore (2):
  - National University Hospital; National University Cancer Institute, Singapore (NCIS), Singapore
  - National Cancer Centre; Medical Oncology, Singapore
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- Spain (3):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - ICO Badalona - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
- Switzerland (4):
  - Universitaetsspital Basel; Onkologie, Basel
  - CHUV; Departement d'Oncologie, Lausanne
  - Kantonsspital St. Gallen; Onkologie/Hämatologie, Sankt Gallen
  - UniversitätsSpital Zürich; Zentrum für Hämatologie und Onkologie, Klinik für Onkologie, Zurich
- Turkey (Türkiye) (4):
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Ankara
  - Ankara Ataturk Chest Diseases Training and Research Hospital, Ankara
  - Ege University School of Medicine; Chest Diseases Department, Izmir
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya
- United Kingdom (3):
  - Barts & London School of Med; Medical Oncology, London
  - Royal Marsden Hospital - London, London
  - Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Saal J, Bald T, Eckstein M, Ralser DJ, Brossart P, Ellinger J, Holzel M, Klumper N. Integration of on-treatment modified Glasgow prognostic score (mGPS) to improve imaging-based prediction of outcomes in patients with non-small cell lung cancer on immune checkpoint inhibition. Lung Cancer. 2024 Mar;189:107505. doi: 10.1016/j.lungcan.2024.107505. Epub 2024 Feb 15. PMID 38367405
- [Derived] Shemesh CS, Chan P, Legrand FA, Shames DS, Das Thakur M, Shi J, Bailey L, Vadhavkar S, He X, Zhang W, Bruno R. Pan-cancer population pharmacokinetics and exposure-safety and -efficacy analyses of atezolizumab in patients with high tumor mutational burden. Pharmacol Res Perspect. 2020 Dec;8(6):e00685. doi: 10.1002/prp2.685. PMID 33241650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Since the primary cut-off date May 8, 2015 one participant in Cohort 1 has moved to Cohort 2 and one participant in Cohort 3 was moved to Cohort 2.
Pre-assignment Details: Screening was performed from Day -28 to Day -1.
Groups:
- Cohort 1: First Line Atezolizumab: Participants received 1200 milligrams (mg) atezolizumab every 3 weeks (Day 1 of 21 day cycle) administered by intravenous (IV) infusion until intolerable toxicity, disease progression or death. Participants in this cohort received no prior chemotherapy in locally advanced or metastatic setting.
- Cohort 2: Second Line Atezolizumab: Participants received 1200 mg atezolizumab every 3 weeks (Day 1 of 21-day cycle) administered by IV infusion until intolerable toxicity, disease progression or death. Participants were permitted to continue treatment after progressive disease, if the following criteria were met: evidence of clinical benefit as assessed by the investigator; absence of symptoms and signs indicating unequivocal progression of disease; no decline in Eastern Cooperative Oncology Group (ECOG) performance status; absence of tumor growth at critical anatomical sites that cannot be managed by protocol-allowed medical interventions; evidence of clinical benefit as assessed by the investigator. Participants in this cohort progressed during or after prior platinum-based chemotherapy in locally advanced or metastatic setting.
- Cohort 3: Third Line and Beyond Atezolizumab: Participants received 1200 mg atezolizumab every 3 weeks ( Day 1 of 21-day cycle) administered by IV infusion until intolerable toxicity, disease progression or death. Participants were permitted to continue treatment after progressive disease, if the following criteria were met: absence of symptoms and signs indicating unequivocal progression of disease; no decline in ECOG performance status; absence of tumor growth at critical anatomical sites that cannot be managed by protocol-allowed medical interventions; evidence of clinical benefit as assessed by the investigator. Participants in this cohort progressed during or after prior platinum-based chemotherapy and at least one additional therapy in locally advanced or metastatic setting.
Period: May 8, 2015 to January 11, 2019
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab
Started | 138 | 269 | 252
Completed | 0 | 0 | 0
Not Completed | 138 | 269 | 252
Not completed — Death | 89 | 193 | 198
Not completed — Lost to Follow-up | 2 | 5 | 8
Not completed — Switched over to commercial Atezolizumab | 1 | 6 | 6
Not completed — Physician Decision | 2 | 3 | 3
Not completed — Protocol Violation | 7 | 4 | 0
Not completed — Study Terminated by Sponsor | 24 | 42 | 23
Not completed — Withdrawal by Subject | 13 | 16 | 14
Period: Baseline to May 8, 2015
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab
Started | 139 | 267 | 253
Completed | 0 | 0 | 0
Not Completed | 139 | 267 | 253
Not completed — Death | 36 | 87 | 100
Not completed — Protocol Violation | 7 | 4 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Unknown Reason | 0 | 1 | 2
Not completed — Withdrawal by Subject | 6 | 9 | 3
Not completed — On Survival Follow-Up | 46 | 83 | 73
Not completed — On Treatment | 43 | 81 | 73
Not completed — Lost to Follow-up | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Efficacy evaluable population included all enrolled participants who received any dose of the study drug (atezolizumab) during the study treatment period.
  Since the primary CSR one patient in Cohort 1 has moved to Cohort 2 and one patient in Cohort 3 was moved to Cohort 2.
Groups:
- Cohort 1: First Line Atezolizumab: Participants received 1200 mg atezolizumab every 3 weeks (Day 1 of 21 day cycle) administered by IV infusion until intolerable toxicity, disease progression or death. Participants in this cohort received no prior chemotherapy in locally advanced or metastatic setting.
- Cohort 2: Second Line Atezolizumab: Participants received 1200 mg atezolizumab every 3 weeks (Day 1 of 21-day cycle) administered by IV infusion until intolerable toxicity, disease progression or death. Participants were permitted to continue treatment after progressive disease, if the following criteria were met: evidence of clinical benefit as assessed by the investigator; absence of symptoms and signs indicating unequivocal progression of disease; no decline in ECOG performance status; absence of tumor growth at critical anatomical sites that cannot be managed by protocol-allowed medical interventions; evidence of clinical benefit as assessed by the investigator. Participants in this cohort progressed during or after prior platinum-based chemotherapy in locally advanced or metastatic setting.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Total
Number analyzed (Participants) | 138 | 269 | 252 | 659
Age, Continuous [Median (Standard Deviation); unit: years] | 66.8 (10.3) | 62.4 (10.2) | 63.6 (9.4) | 63.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 104 | 100 | 272
  Male | 70 | 165 | 152 | 387

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Objective Response (ORR) Per Response Evaluation Criteria In Solid Tumors (RECIST) Version (v) 1.1 as Assessed by Independent Review Facility (IRF)
Description: ORR was the percentage of participants whose confirmed best overall response was either a Partial Response (PR) or a Complete Response (CR) based upon the IRF assessment per RECIST v1.1. CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm); PR:greater than (>) or equal to (=) 30 percent (%) decrease from baseline in sum of diameters of target lesions, non-progressive disease (PD) non-target lesions and no new lesions. Results were reported by line of therapy and programmed death-ligand 1 (PD-L1) Expression Subgroup (tumor cell [TC]3 [TC3] or tumor-infiltrating immune cell [IC] 3 [IC3], TC3 or IC2/3, TC2/3 or IC2/3).
Time Frame: Screening, Every 6 weeks (± 3 days) for 12 months following Cycle 1, Day 1 and every 9 weeks (± 1 week) thereafter until disease progression, intolerable toxicity or death until data cut-off on 28 May 2015 (Up to 16 months)
Population: Efficacy evaluable population; Number (n) equals (=) number of participants analyzed within the specified group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohorts 2 + 3: This sub-group included participants from cohorts 2 and 3. All participants who were treated and had evaluable pharmacokinetic samples were included in this group.
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3 Responders: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 Responders | 26.2 [16.0 to 38.5] | 23.8 [16.5 to 32.3] | 27.0 [19.1 to 36.0] | 25.35 [19.9 to 31.4]
  TC3 or IC2/3 Responders: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 Responders | 21.1 [14.3 to 29.4] | 17.4 [12.9 to 22.7] | 18.2 [13.5 to 23.8] | 17.8 [14.5 to 21.5]
  TC2/3 or IC2/3 Responders | 19.4 [13.2 to 27.0] | 17.2 [12.9 to 22.3] | 17.4 [12.9 to 22.6] | 17.3 [14.2 to 20.8]

2. Secondary Outcome: Percentage of Participants Achieving Objective Response Per RECIST v1.1 as Assessed by the Investigator (INV)
Description: ORR was the percentage of participants whose confirmed best overall response was either a PR or a CR based upon the Investigator assessment per RECIST v1.1. CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10mm; PR: > or = 30 % decrease from baseline in sum of diameters of target lesions, non-PD non-target lesions and no new lesions. Results were reported by line of therapy (reporting arms) and PD-L1 Expression Subgroup (TC3 or IC3, TC3 or IC2/3, TC2/3 or IC2/3).
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3 Responders: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 Responders | 30.8 [19.9 to 43.5] | 24.6 [17.3 to 33.2] | 28.7 [20.7 to 37.9] | 26.6 [21.1 to 32.7]
  TC3 or IC2/3 Responders: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 Responders | 24.4 [17.1 to 33.0] | 19.4 [14.7 to 24.9] | 19.1 [14.3 to 24.7] | 19.3 [15.8 to 23.1]
  TC2/3 or IC2/3 Responders (n= 139, 267, 253, 520) | 22.3 [15.7 to 30.1] | 18.7 [14.2 to 23.9] | 18.2 [13.6 to 23.5] | 18.5 [15.2 to 22.1]

3. Secondary Outcome: Percentage of Participants Achieving Objective Response Per Modified RECIST as Assessed by the INV
Description: ORR was the percentage of participants whose confirmed best overall response was either a PR or a CR based upon the Investigator assessment per modified RECIST. CR: disappearance of all target lesions. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10mm; PR: At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions, taking as reference the baseline sum of diameters, in the absence of CR. Results were reported by line of therapy (reporting arms) and PD-L1 Expression Subgroup (TC3 or IC3, TC3 or IC2/3, TC2/3 or IC2/3).
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n= number of participants analyzed within the specified group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3 Responders: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 Responders | 20.0 [11.1 to 31.8] | 27.0 [19.4 to 35.8] | 30.4 [22.2 to 39.7] | 28.7 [23.0 to 34.9]
  TC3 or IC2/3 Responders: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 Responders | 16.3 [10.2 to 24.0] | 21.9 [16.9 to 27.5] | 20.8 [15.8 to 26.5] | 21.3 [17.8 to 25.3]
  TC2/3 or IC2/3 Responders | 15.8 [10.2 to 23.0] | 21.0 [16.3 to 26.4] | 19.8 [15.0 to 25.2] | 20.4 [17.0 to 24.1]

4. Secondary Outcome: Duration of Response (DOR) Assessed by IRF Per RECIST v1.1
Description: DOR is interval between date of first occurrence of a CR or PR that is subsequently confirmed (whichever status is recorded first) and the first date that PD or death is documented, whichever occurs first as measured by RECIST v1.1. CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10mm; PR: > or = 30 % decrease from baseline in sum of diameters of target lesions, non-PD non-target lesions and no new lesions; PD: one or more of the following: at least 20% increase from nadir in sum of diameters of target lesions (with an absolute increase of at least 5mm), appearance of new lesions, and/or unequivocal progression of non-target lesions. DOR was assessed by Kaplan-Meier estimates. Results were reported by line of therapy (reporting arms) and PD-L1 Expression Subgroup (TC3 or IC3, TC3 or IC2/3, TC2/3 or IC2/3).
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group. Number of participants analyzed = overall number of participants who were evaluable for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 27 | 46 | 44 | 90
months
  TC3 or IC3 DOR: number analyzed (Participants) | 17 | 29 | 31 | 60
  TC3 or IC3 DOR | NA [5.8 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [4.9 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 7.2 [5.6 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 7.2 [5.7 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  TC3 or IC2/3 DOR: number analyzed (Participants) | 26 | 43 | 43 | 86
  TC3 or IC2/3 DOR | 8.5 [5.6 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.4 [6.9 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.4 [5.7 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.4 [6.9 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  TC2/3 or IC2/3 DOR | 8.5 [5.6 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.4 [6.9 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.4 [5.7 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.4 [6.9 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.

5. Secondary Outcome: DOR as Assessed by INV Per RECIST v1.1
Description: DOR is interval between date of the first occurrence of a CR or PR that is subsequently confirmed (whichever status is recorded first) and first date that PD or death is documented, whichever occurs first as measured by RECIST v1.1. CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10mm; PR: > or = 30 % decrease from baseline in sum of diameters of target lesions, non-PD non-target lesions and no new lesions; PD: one or more of the following: at least 20% increase from nadir in sum of diameters of target lesions (with an absolute increase of at least 5mm), appearance of new lesions, and/or unequivocal progression of non-target lesions. DOR was assessed by Kaplan-Meier estimates. Results were reported by line of therapy (reporting arms) and PD-L1 Expression Subgroup (TC3 or IC3, TC3 or IC2/3, TC2/3 or IC2/3).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 81 | 128 | 124 | 252
months
  TC3 or IC3 DOR: number analyzed (Participants) | 20 | 30 | 33 | 63
  TC3 or IC3 DOR | 8.5 [5.6 to 8.5] | NA [8.1 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.4 [6.4 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [7.4 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  TC3 or IC2/3 DOR: number analyzed (Participants) | 30 | 48 | 45 | 93
  TC3 or IC2/3 DOR | 8.5 [8.5 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.3 [7.0 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [8.3 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  TC2/3 or IC2/3 DOR: number analyzed (Participants) | 31 | 50 | 46 | 96
  TC2/3 or IC2/3 DOR | NA [8.5 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.3 [7.0 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [8.3 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.

6. Secondary Outcome: DOR as Assessed by INV Per Modified RECIST
Description: DOR is the interval between the date of the first occurrence of a CR or PR that is subsequently confirmed (whichever status is recorded first) and the first date that PD or death is documented, whichever occurs first as measured by modified RECIST. CR: disappearance of all target lesions. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10mm; PR: at least a 30% decrease in the sum of the diameters of all target and all new measurable lesions, taking as reference the baseline sum of diameters, in the absence of CR; PD: one or more of the following: at least 20% increase from nadir in the sum of diameters of existing and/or new target lesions (with an absolute increase of at least 5mm). DOR was assessed by Kaplan-Meier estimates. Results were reported by line of therapy (reporting arms) and PD-L1 Expression Subgroup (TC3 or IC3, TC3 or IC2/3, TC2/3 or IC2/3).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 55 | 143 | 134 | 277
months
  TC3 or IC3 DOR: number analyzed (Participants) | 13 | 33 | 35 | 68
  TC3 or IC3 DOR | NA [4.4 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [8.1 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [7.4 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [8.1 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  TC3 or IC2/3 DOR: number analyzed (Participants) | 20 | 54 | 49 | 103
  TC3 or IC2/3 DOR | NA [NA to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [7.4 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  TC2/3 or IC2/3 DOR: number analyzed (Participants) | 22 | 56 | 50 | 106
  TC2/3 or IC2/3 DOR | NA [4.5 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [7.4 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.

7. Secondary Outcome: Progression Free Survival (PFS) as Assessed by IRF Per RECIST v1.1
Description: PFS is the interval between the first dose of atezolizumab and date of disease progression or death due to any cause, whichever occurred first as measured by RECIST v1.1. PD is defined as one or more of the following: at least 20% increase from nadir in the sum of diameters of target lesions (with an absolute increase of at least 5mm), appearance of new lesions, and/or unequivocal progression of non-target lesions. PFS was assessed by Kaplan-Meier estimates.
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
months
  TC3 or IC3 PFS: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 PFS | 5.5 [2.7 to 8.3] | 4.1 [1.8 to 5.5] | 4.2 [2.8 to 5.6] | 4.1 [2.8 to 5.4]
  TC3 or IC2/3 PFS: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 PFS | 5.6 [3.3 to 8.3] | 2.8 [1.5 to 4.0] | 2.8 [2.7 to 4.0] | 2.8 [2.7 to 3.0]
  TC2/3 or IC2/3 PFS | 5.5 [3.0 to 6.9] | 2.8 [1.5 to 3.5] | 2.8 [2.7 to 3.7] | 2.8 [2.7 to 2.9]

8. Secondary Outcome: PFS as Assessed by INV Per RECIST v1.1
Description: PFS is the interval between the first dose of atezolizumab and date of disease progression or death due to any cause, whichever occurred first as measured by RECIST v1.1. PD: one or more of the following: at least 20% increase from nadir in the sum of diameters of target lesions (with an absolute increase of at least 5mm), appearance of new lesions, and/or unequivocal progression of non-target lesions. PFS was assessed by Kaplan-Meier estimates.
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
months
  TC3 or IC3 PFS: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 PFS | 7.1 [4.9 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 4.1 [2.7 to 6.5] | 4.2 [3.0 to 6.2] | 4.2 [2.9 to 5.6]
  TC3 or IC2/3 PFS: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 PFS | 7.6 [5.9 to 9.9] | 3.0 [2.7 to 4.2] | 3.5 [2.8 to 4.2] | 3.2 [2.8 to 4.1]
  TC2/3 or IC2/3 PFS | 7.1 [5.6 to 8.4] | 2.8 [2.6 to 4.1] | 3.0 [2.8 to 4.1] | 3.0 [2.8 to 4.1]

9. Secondary Outcome: PFS as Assessed by INV Per Modified RECIST
Description: PFS is the interval between the first dose of atezolizumab and date of disease progression or death due to any cause, whichever occurred first as measured by modified RECIST. PD: at least 20% increase from nadir in the sum of diameters of new and/or existing target lesions (with an absolute increase of at least 5mm). PFS was assessed by Kaplan-Meier estimates.
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
months
  TC3 or IC3 PFS: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 PFS | 7.1 [4.7 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 5.7 [4.1 to 8.4] | 6.3 [4.1 to 8.1] | 5.8 [4.3 to 7.1]
  TC3 or IC2/3 PFS: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 PFS | 7.9 [5.7 to 10.0] | 4.5 [4.0 to 6.0] | 4.9 [4.1 to 6.8] | 4.6 [4.1 to 5.7]
  TC2/3 or IC2/3 PFS | 7.6 [5.6 to 9.9] | 4.2 [3.9 to 5.7] | 4.6 [4.1 to 6.3] | 4.4 [4.1 to 5.5]

10. Secondary Outcome: Overall Survival : Percentage of Participants Without Event (Death)
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 | 70.8 | 70.5 | 67.0 | 68.8
  TC3 or IC2/3: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 | 75.6 | 69.2 | 60.6 | 65.0
  TC2/3 or IC2/3 | 74.1 | 67.4 | 60.5 | 64.0

11. Secondary Outcome: Overall Survival : Median Time to Event (Death)
Description: Overall survival is measured as interval between the first dose of atezolizumab and date of death from any cause.
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
months
  TC3 or IC3: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 | NA [10.4 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [10.6 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [12.1 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  TC3 or IC2/3: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 | 14.0 [14.0 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [12.1 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [8.4 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [12.1 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  TC2/3 or IC2/3 | 14.0 [14.0 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [11.2 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [8.4 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [11.2 to NA] — Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.

12. Secondary Outcome: Percentage of Participants Without an Event (Death) at 6 Months
Time Frame: Month 6
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 | 79.2 [69.1 to 89.3] | 79.7 [72.5 to 87.0] | 75.1 [67.1 to 83.1] | 77.4 [72.0 to 82.8]
  TC3 or IC2/3: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 | 83.9 [77.2 to 90.5] | 78.1 [72.8 to 83.4] | 71.0 [65.2 to 76.9] | 74.6 [70.6 to 78.5]
  TC2/3 or IC2/3 | 81.7 [75.1 to 88.4] | 76.2 [71.0 to 81.5] | 70.5 [64.9 to 76.2] | 73.4 [69.5 to 77.3]

13. Secondary Outcome: Percentage of Participants Without an Event (Death) at 12 Months
Time Frame: Month 12
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 | 58.6 [40.7 to 76.5] | 61.5 [49.0 to 74.0] | 62.6 [52.8 to 72.5] | 61.3 [52.7 to 69.8]
  TC3 or IC2/3: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 | 67.1 [55.7 to 78.4] | 59.3 [50.5 to 68.1] | 54.9 [47.7 to 62.2] | 56.5 [50.6 to 62.5]
  TC2/3 or IC2/3 | 65.0 [54.0 to 76.1] | 57.2 [48.6 to 65.7] | 54.4 [47.3 to 61.5] | 55.3 [49.5 to 61.1]

14. Secondary Outcome: PFS: Percentage of Participants Alive and Progression Free at 6 Months
Description: PD is defined as one or more of the following: at least 20% increase from nadir in the sum of diameters of target lesions (with an absolute increase of at least 5mm), appearance of new lesions, and/or unequivocal progression of non-target lesions.
Time Frame: Month 6
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 | 57.4 [44.7 to 70.1] | 41.3 [32.3 to 50.4] | 42.1 [33.1 to 51.2] | 41.8 [35.4 to 48.2]
  TC3 or IC2/3: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 | 58.6 [49.5 to 67.8] | 36.1 [29.9 to 42.2] | 35.8 [29.6 to 41.9] | 35.9 [31.6 to 40.3]
  TC2/3 or IC2/3 | 56.4 [47.8 to 65.1] | 34.8 [29.0 to 40.7] | 34.7 [28.7 to 40.6] | 34.8 [30.6 to 38.9]

15. Secondary Outcome: PFS: Percentage of Participants Alive and Progression Free at 12 Months
Description: as for outcome 14
Time Frame: Month 12
Population: Efficacy evaluable population; n = number of participants analyzed within the specified group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 | 33.1 [14.9 to 51.3] | 27.8 [17.6 to 37.9] | 16.1 [3.8 to 28.5] | 23.1 [15.4 to 30.8]
  TC3 or IC2/3: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 | 29.0 [13.1 to 45.0] | 22.7 [16.1 to 29.3] | 15.1 [8.3 to 21.8] | 19.1 [14.4 to 23.8]
  TC2/3 or IC2/3 | 26.9 [12.1 to 41.7] | 21.8 [15.5 to 28.1] | 14.7 [8.1 to 21.3] | 18.5 [14.0 to 23.1]

16. Secondary Outcome: Time in Response (TIR) as Assessed by INV Per RECIST v1.1
Description: TIR is interval between date of first occurrence of a CR or PR that is subsequently confirmed (whichever status is recorded first) and first date that PD or death is documented, whichever occurs first as measured by RECIST v1.1. For responders, TIR was the same as DOR; for non-responders, TIR was considered as an event and defined as the date of first treatment plus one day. TIR was assessed by Kaplan-Meier estimates.
Time Frame: as for outcome 1
Population: Efficacy evaluable population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
months | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events.

17. Secondary Outcome: TIR as Assessed by INV Per Modified RECIST
Description: TIR is interval between date of first occurrence of a CR or PR that is subsequently confirmed (whichever status is recorded first) and first date that PD or death is documented, whichever occurs first as measured by modified RECIST. For responders, TIR was the same as DOR; for non-responders, TIR was considered as an event and defined as the date of first treatment plus one day. TIR was assessed by Kaplan-Meier estimates.
Time Frame: as for outcome 1
Population: Efficacy evaluable population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
months | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events.

18. Secondary Outcome: TIR as Assessed by IRF Per RECIST v1.1
Description: as for outcome 16
Time Frame: as for outcome 1
Population: Efficacy evaluable population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
months | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 0.033 [NA to NA] — Median reported is the censored value, confidence interval not estimable by Brookmeyer and Crowley method due to insufficient observed events.

19. Secondary Outcome: Atezolizumab Serum Concentrations
Description: Serum concentrations were determined for all participants after administration of atezolizumab up to Cycle 8. Time (T) = time from first dose in days.
Time Frame: Pre-dose (hour 0) and 0.5 hours post dose on Cycle 1 Day 1 (Cycle length = 21days), Cycle 1 Days 2, 4, 8, 15, and 21, Cycle 2 Day 21, Cycle 3 Day 21, Cycle 7 Day 21
Population: Pharmacokinetic evaluable population; n = number of participants analyzed for the specified time point.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Groups:
- Pharmacokinetic Evaluable Population: Participants received 1200 milligrams (mg) atezolizumab every 3 weeks (Day 1 of 21 day cycle) administered by intravenous (IV) infusion until intolerable toxicity, disease progression or death. All participants who were treated and had evaluable pharmacokinetic samples were included in this group.
Arm/Group | Pharmacokinetic Evaluable Population
Number analyzed (Participants) | 646
micrograms per milliliter (μg/mL)
  Cycle 1 Day 1 T=0 | 0.285 (4.35)
  Cycle 1 Day 1 T=0.021 | 429.0 (218)
  Cycle 1 Day 2 T=1: number analyzed (Participants) | 47
  Cycle 1 Day 2 T=1 | 299.0 (65.3)
  Cycle 1 Day 4 T=3: number analyzed (Participants) | 44
  Cycle 1 Day 4 T=3 | 220.0 (48.4)
  Cycle 1 Day 8 T=7: number analyzed (Participants) | 38
  Cycle 1 Day 8 T=7 | 155.0 (35.4)
  Cycle 1 Day 15 T=14: number analyzed (Participants) | 36
  Cycle 1 Day 15 T=14 | 106.0 (32.1)
  Cycle 1 Day 21 T=21: number analyzed (Participants) | 596
  Cycle 1 Day 21 T=21 | 87.8 (41.7)
  Cycle 2 Day 21 T=42: number analyzed (Participants) | 518
  Cycle 2 Day 21 T=42 | 134.0 (57.2)
  Cycle 3 Day 21 T=63: number analyzed (Participants) | 467
  Cycle 3 Day 21 T=63 | 163.0 (70.7)
  Cycle 7 Day 21 T=147: number analyzed (Participants) | 275
  Cycle 7 Day 21 T=147 | 212.0 (88.5)

20. Secondary Outcome: Percentage of Participants With Positive Anti-Therapeutic Antibody (Anti-Atezolizumab Antibody) Status
Description: Anti-therapeutic antibodies is a measurement to explore the potential relationship of immunogenicity response with pharmacokinetics, safety and efficacy.
Time Frame: Baseline, post-baseline (up to 16 months)
Population: Efficacy evaluable population; n = number of participants analyzed at the specified time point. Number of participants analyzed = number participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 135 | 257 | 247 | 504
percentage of participants
  Baseline | 7.4 | 3.5 | 6.1 | 4.8
  Post-Baseline: number analyzed (Participants) | 133 | 253 | 238 | 491
  Post-Baseline | 45.1 | 36.0 | 37.4 | 36.7

21. Secondary Outcome: Percentage of Participants With Event (Disease Progression or Death) as Assessed by IRF Per RECIST v1.1
Description: PD was defined as one or more of the following: at least 20% increase from nadir in the sum of diameters of target lesions (with an absolute increase of at least 5 mm), appearance of new lesions, and/or unequivocal progression of non-target lesions.
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 | 58.5 | 68.0 | 73.0 | 70.5
  TC3 or IC2/3: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 | 61.8 | 73.7 | 79.2 | 76.4
  TC2/3 or IC2/3 | 63.3 | 75.3 | 79.1 | 77.1

22. Secondary Outcome: Percentage of Participants With Event (Disease Progression or Death) as Assessed by INV Per RECIST v1.1
Description: as for outcome 21
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 | 50.8 | 63.1 | 68.7 | 65.8
  TC3 or IC2/3: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 | 50.4 | 68.8 | 74.6 | 71.6
  TC2/3 or IC2/3 | 52.5 | 70.0 | 74.7 | 72.3

23. Secondary Outcome: Percentage of Participants With Event (Disease Progression or Death) as Assessed by INV Per Modified RECIST v1.1
Description: PD was defined as at least 20% increase from nadir in the sum of diameters of new and/or existing target lesions (with an absolute increase of at least 5 mm).
Time Frame: as for outcome 1
Population: Efficacy evaluable population; n = number of participants analyzed at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab | Cohorts 2 + 3
Number analyzed (Participants) | 139 | 267 | 253 | 520
percentage of participants
  TC3 or IC3: number analyzed (Participants) | 65 | 122 | 115 | 237
  TC3 or IC3 | 36.9 | 56.6 | 60.0 | 58.2
  TC3 or IC2/3: number analyzed (Participants) | 123 | 247 | 236 | 483
  TC3 or IC2/3 | 38.2 | 61.5 | 66.1 | 63.8
  TC2/3 or IC2/3 | 39.6 | 62.9 | 66.4 | 64.6

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of Screening until 30 days after the final follow-up visit until data cut-off on 11 January 2019 (Up to 60 months)
Arm/Group | Cohort 1: First Line Atezolizumab | Cohort 2: Second Line Atezolizumab | Cohort 3: Third Line and Beyond Atezolizumab
All-Cause Mortality (participants affected / at risk) | 89/138 | 193/269 | 198/252
Serious Adverse Events (participants affected / at risk) | 47/138 | 117/269 | 113/252
Other Adverse Events (participants affected / at risk) | 116/138 | 229/269 | 229/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: First Line Atezolizumab (N=138) | Cohort 2: Second Line Atezolizumab (N=269) | Cohort 3: Third Line and Beyond Atezolizumab (N=252)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4)
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENITIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
CARDIAC TAMPONADE (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (5) | 2 (3)
OESOPHAGEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 4 (7) | 3 (3)
ASTHENIA (General disorders) | 1 (1) | 1 (1) | 3 (3)
CHEST PAIN (General disorders) | 0 (0) | 2 (2) | 2 (2)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 0 (0) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERTHERMIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1) | 0 (0)
MALAISE (General disorders) | 0 (0) | 2 (3) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 9 (9) | 8 (8)
SUDDEN DEATH (General disorders) | 0 (0) | 1 (1) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC HAEMORRHAGE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATOMEGALY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
CATHETER SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
EMPYEMA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
FEBRILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 1 (1) | 3 (4) | 2 (2)
MEDIASTINITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 6 (6) | 15 (19) | 16 (18)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
VESTIBULAR NEURONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (3) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TRAUMATIC HAEMOTHORAX (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 6 (7) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC COMPRESSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LYMPHANGIOSIS CARCINOMATOSA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PLEURAL MESOTHELIOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
APRAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
FACIAL PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MOTOR DYSFUNCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MYELOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PARAPLEGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
RENAL INFARCT (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
SCROTAL PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
ACQUIRED TRACHEO-OESOPHAGEAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
BRONCHIAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6) | 11 (12)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (6) | 4 (4)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
LARYNGEAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 6 (7)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
TRACHEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
ALCOHOL DETOXIFICATION (Surgical and medical procedures) | 0 (0) | 1 (3) | 0 (0)
DRUG DETOXIFICATION (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
EMBOLISM (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
INTERNAL HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
PHLEBITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: First Line Atezolizumab (N=138) | Cohort 2: Second Line Atezolizumab (N=269) | Cohort 3: Third Line and Beyond Atezolizumab (N=252)
ANAEMIA (Blood and lymphatic system disorders) | 17 (33) | 31 (54) | 22 (41)
HYPOTHYROIDISM (Endocrine disorders) | 8 (10) | 15 (16) | 10 (16)
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 (12) | 22 (27) | 18 (24)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (7) | 6 (7) | 15 (18)
CONSTIPATION (Gastrointestinal disorders) | 19 (27) | 47 (57) | 45 (57)
DIARRHOEA (Gastrointestinal disorders) | 29 (51) | 64 (99) | 47 (93)
DRY MOUTH (Gastrointestinal disorders) | 10 (11) | 18 (19) | 10 (12)
NAUSEA (Gastrointestinal disorders) | 29 (48) | 69 (99) | 60 (90)
VOMITING (Gastrointestinal disorders) | 21 (32) | 41 (54) | 36 (53)
ASTHENIA (General disorders) | 13 (19) | 27 (49) | 40 (87)
CHEST PAIN (General disorders) | 5 (7) | 24 (30) | 26 (30)
CHILLS (General disorders) | 5 (5) | 15 (18) | 14 (15)
FATIGUE (General disorders) | 52 (70) | 85 (145) | 92 (142)
INFLUENZA LIKE ILLNESS (General disorders) | 13 (17) | 24 (30) | 13 (18)
MALAISE (General disorders) | 9 (10) | 8 (10) | 9 (9)
MUCOSAL INFLAMMATION (General disorders) | 7 (7) | 11 (13) | 10 (17)
OEDEMA PERIPHERAL (General disorders) | 10 (11) | 22 (32) | 22 (26)
PAIN (General disorders) | 11 (17) | 15 (19) | 11 (12)
PYREXIA (General disorders) | 20 (24) | 47 (63) | 45 (60)
LUNG INFECTION (Infections and infestations) | 7 (7) | 3 (3) | 11 (13)
NASOPHARYNGITIS (Infections and infestations) | 14 (16) | 11 (18) | 18 (25)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 16 (18) | 26 (45) | 20 (27)
URINARY TRACT INFECTION (Infections and infestations) | 8 (14) | 18 (29) | 14 (19)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 14 (17) | 12 (17)
BLOOD CREATININE INCREASED (Investigations) | 4 (4) | 16 (22) | 6 (7)
WEIGHT DECREASED (Investigations) | 7 (7) | 22 (28) | 29 (35)
DECREASED APPETITE (Metabolism and nutrition disorders) | 34 (40) | 55 (70) | 74 (106)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 (13) | 6 (6) | 9 (11)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 19 (29) | 41 (70) | 37 (58)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 22 (28) | 35 (51) | 35 (46)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 9 (10) | 10 (11) | 5 (5)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 9 (9) | 15 (18) | 14 (19)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7 (8) | 23 (25) | 27 (41)
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 (7) | 19 (28) | 16 (18)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 10 (12) | 12 (15) | 14 (17)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 15 (23) | 28 (39) | 25 (38)
DIZZINESS (Nervous system disorders) | 7 (9) | 27 (39) | 21 (25)
HEADACHE (Nervous system disorders) | 19 (25) | 22 (33) | 35 (43)
ANXIETY (Psychiatric disorders) | 5 (5) | 18 (23) | 17 (19)
DEPRESSION (Psychiatric disorders) | 8 (9) | 12 (14) | 8 (10)
INSOMNIA (Psychiatric disorders) | 12 (12) | 20 (23) | 21 (25)
COUGH (Respiratory, thoracic and mediastinal disorders) | 44 (75) | 66 (94) | 81 (117)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 42 (69) | 49 (67) | 69 (106)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 17 (20) | 15 (27)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 4 (4) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (17) | 23 (26) | 15 (24)
DRY SKIN (Skin and subcutaneous tissue disorders) | 14 (16) | 19 (20) | 16 (20)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 5 (5) | 17 (19) | 7 (10)
PRURITUS (Skin and subcutaneous tissue disorders) | 20 (29) | 43 (64) | 36 (55)
RASH (Skin and subcutaneous tissue disorders) | 21 (33) | 34 (47) | 29 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.